CLINICAL TRIAL: NCT03387436
Title: Treatment as Usual vs. Additional Collaborative Advance Care Planning to Improve Quality of Life for Palliative Cancer Patients: a Randomized Controlled Trial
Brief Title: The "Hand-in-Hand Study": Improvement of Quality of Life in Palliative Cancer Patients Through Collaborative Advance Care Planning
Acronym: COLAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PD. Dr. med. Carola Seifart (Other)
Collaborators: Philipps University Marburg (Other); German Federal Ministry of Education and Research (Other Government); Department of Clinical Psychology and Psychotherapy (Unknown)
Responsible Party: Sponsor-Investigator, PD. Dr. med. Carola Seifart, Sponsor-Investigator, Philipps University Marburg
Organization: Philipps University Marburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 01GY1708; 01GY1708 (Other Grant/Funding Number: Federal Ministry of Education and Research)
Record Dates: First submitted 2017-12-04; First posted 2018-01-02 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Advanced Cancer; Neoplasms; End Stage Cancer
Keywords: Palliative care; Advance care planning; psychological intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be allocated randomly to three arms:
  1. palliative treatment as usual (TAU)
  2. sham-intervention + (TAU)
  3. study-intervention + (TAU)
  Stratification will be carried out for sex, and availability of a care giver.
Who Masked: Investigator, Outcomes Assessor
Masking Description: As in most psychological interventions, care providers (psychologists) can not be blinded, because they are delivering the intervention.
  Patients only know if they are in one of the intervention groups or in TAU. All other study personnel will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.) Treatment as usual (TAU) (No Intervention): Patients assigned to this arm will receive palliative treatment as usual.
- 2.) Sham-Intervention (Sham Comparator): Patients assigned to this arm will receive an sham intervention with unspecific supportive therapy (i.e. listening, empathy etc., but no specific intervention rationale) and palliative treatment as usual.
  Interventions: Behavioral: Sham-Intervention
- 3.) Study-Intervention (Experimental): Patients assigned to this arm will receive the study-intervention and palliative treatment as usual.
  Interventions: Behavioral: Study-Intervention

INTERVENTIONS:
Behavioral: Sham-Intervention — The sham intervention does not target the specific topics of the study intervention group (i.e. no special focus an ACP or end of life communication). Supportive therapy uses common factors of psychotherapy such as elicitation of affect, reflective listening, and feeling understood, but provides no explicit theoretical formulation to the patient. The therapist tries to elicit and validate the patients' affect for instance on the realization that there is no curative treatment option. Supportive therapy has been used as an unspecific control condition in several studies (Cohen et al. 2011; Markowitz et al. 1998). Patients of the sham intervention will be informed about the benefits of advance directives in general.
  Arms: 2.) Sham-Intervention
Behavioral: Study-Intervention — The design of the study-intervention was influenced by dignity therapy (Chochinov et al. 2005), the End-of-life-Review (Ando et al. 2010) and barriers concerning participation of ACP identified by research (Bollig et al. 2017; Gjerberg et al. 2015). It is the goal of the study-intervention to enhance communication about death related topics of patients and their relatives/caregivers.
  Our study intervention extends over six therapeutic sessions. The length of each session will be adjusted to the patients physical condition, it should not exceed 45 minutes in total.
  In the first four sessions, patients and relatives will be informed about the relevance of ACP. Potential barriers for an efficient patient-caregiver communication and ACP are discussed. The intervention focuses on encouraging end-of-life communication and on jointly modifying barriers to EOL communication.
  The fifth and sixth session focus on ACP based on the standardised concept of "beizeiten begleiten".
  Arms: 3.) Study-Intervention

SUMMARY:
This study evaluates the effect of a collaborative advance care planning intervention on the quality of life in palliative oncological patients. Research indicates, that talking about wishes for end of life care and death, may improve the quality of life, but can be difficult for involved parties.

The intervention especially developed for this study trys to reduce psychosocial barriers that make conversations about these topics difficult. The study will measure the effect of the intervention on patients and caregivers quality of life.

The study will give additional information about implementation of advance care planning interventions in different care settings in a complex health care systems.

DETAILED DESCRIPTION:
A high quality of end of life care and a "good death" as part of an improved patient centered care at the end of life have become important goals of palliative care. To achieve these goals, patient's preferences for end of life (EOL) care need to be known.

This study (randomized controlled trial) will evaluate effectiveness of a new type of advance care planning (ACP) intervention in different palliative care settings in Germany. The study addresses a new concept of ACP called collaborative advance care planning (cACP). This new concept is focusing on psychosocial barriers of patients and caregivers in addition to a standardized ACP process in order to reduce distress of patients and care-givers and enhance the chance of successful ACP-implementation. The main research questions are: a) Can cACP improve quality of life in palliative patients and caregivers?, b) Does cACP reduce distress in patients and caregivers and enhance consistency of end-of-life care? and c) Does cACP improve quality of end of life care and reduce utilization of health care resources? The investigators will try to answer theses research questions through a so called "randomized controlled trial" methodology. Admissible palliative cancer patients who are willing to participate in the trial will be randomly assigned to three groups. The first group will receive treatment as usual for palliative care patients. The second group will receive treatment as usual and an unspecific psychological intervention (sham-intervention). The third group will receive treatment as usual and the intervention designed for this trial. Both interventions will be equally long in duration and will be delivered by the same psychologists.

The primary outcome is the quality of life at 16 weeks measured by the internationally recognized "Functional Assessment of Cancer - General Version (FACT-G)" questionnaire. Secondary endpoints include measurements of the development of QoL over time, distress, depression, and the quantity of advance directives in the different groups.

Patients will be recruited in four different recruiting sites: a palliative care ward in an university hospital, an oncologists office, a rehabilitation clinic, and an outpatient palliative care network.

The study will recruit 90 patients in every group, 270 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years
* Patient with advance cancer in palliative setting
* positive surprise question: the physician will not be surprised, if the patient died in the next 12 month
* Patient is willing to take part in the study

Exclusion Criteria:

* Patients life expectancy below 3 month (estimated by physician)
* Patients ECOG-status is > 3
* Patient is not able to speak German
* Patient is incapacitated to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
The Functional Assessment of Cancer Therapy scale (FACT-G; Cella, Tulsky, Gray, et al., 1993) | 60 weeks; Baseline, 8 weeks (after randomisation: a.r.), 16 weeks (a. r.); every two month for the following 8 month or till death (if occuring within one year after randomisation)
  Quality of life (QOL). Self-rating measurement; four subscales: physical well-being (7-items, score range 0-28), social/ family well-being (7-items, score range 0-28), emotional well being (6-items, score range 0-24) and functional well being (7-items, score range 0-28), one total score (sum of the four subscale scores; score range of 0-108). Higher subscale and total scores indicate better QoL.

SECONDARY OUTCOMES:
12-Item Short Form Health Survey (SF-12; Ware, Kosinski, Keller, 1996) | 60 weeks; Baseline, 8 weeks (after randomisation: a.r.), 16 weeks (a. r.); every two month for the following 8 month or till death (if occuring within one year after randomisation)
  QOL of patients. Two subscales of health related quality of life (QOL): physical health and mental health (score range:0-100). Higher scores indicate better QoL.
Functional assessment of chronic illness therapy - palliative care- 14 items (FACIT-Pal-14; Zeng et al. 2014) | 60 weeks; Baseline, 8 weeks (after randomisation: a.r.), 16 weeks (a. r.); every two month for the following 8 months or till death (if occuring one year after randomisation)
  QoL of palliative care patients. A higher score indicate better QoL.
National Comprehensive Cancer Network Distress Thermometer (Mehnert et al. 2006) | 16 weeks; Baseline, 8 weeks (after randomisation: a.r.), 16 weeks (a. r.)
  scale from 0 to 10 assessing overall psycho social distress, was specifically developed for oncological patients.
Peace, Equanimity, and Acceptance in the Cancer Experience (PEACE-Scale, Mack et al. 2008) | 16 weeks; Baseline, 8 weeks (after randomisation: a.r.), 16 weeks (a. r.)
  The scale was developed to assess the acceptance of the disease and the inner peace of patients.
  12 items, two subscales: inner acceptance of disease (score 0-20 high number indicating high acceptance), inner conflict with disease (score 0-28 high score indicating more conflict)
Barriers of communication (patients) | 8 weeks; Baseline, 8 weeks (after randomisation: a.r.)
  This self developed questionnaire will try to assess the barriers of communication of patients and caregivers concerning topics like end of life care and death.
  25 items, 6 point likert scale. High score indicating low barriers of communication (some reverse scored items). The scale will be validated in the study.
Patient Health Questionnaire (PHQ-9; Kroenke et al. 2001) | 16 weeks; Baseline, 8 weeks (after randomisation: a.r.), 16 weeks (a. r.)
  Assesses severe symptoms of depression based on criteria by the DSM IV. 9 items, sumscore (0-27), a high sumscore indicates a high level of depression
Expectations about treatment of patients (self-developed, visual analogues scale) | 16 weeks; Baseline, 16 weeks (a. r.)
  These three self-developed items assess descriptive 1. the expectations patients have towards their cancer therapy (e.g. prolonging of life, improvement of QoL) and 2. the importance of prolonging of life & improvement of QoL (two visual analogues scales)
Existence of ACP directive | 60 weeks; Baseline, 8 weeks (after randomisation: a.r.), 16 weeks (a. r.); 1 year (a.r.) or after death (if occuring one year a. r.)
  Patients will be asked, if they have completed and advance healthcare directive or took part in an ACP-process. Purely descriptive (Advance directive yes vs. no)
Caregiver Quality of Life Index - Cancer Scale (CQOLC; Weitzner et al., 1999) | 60 weeks; Baseline, 8 weeks (after randomisation: a.r.), 16 weeks (a. r.); 1 year (a.r.) or after death of patient (if occuring one year a. r.)
  Assessment of cancer caregivers QoL and has been validated in curative and palliative settings.
  34 items, 5 point likert scale, high score indicating low QoL (some items reverse scoreed)
12-Item Short Form Health Survey (SF-12; Ware, Kosinski & Keller,1996) | 60 weeks; Baseline, 8 weeks (after randomisation: a.r.), 16 weeks (a. r.); 1 year (a.r.) or after death of patient (if occuring one year a. r.)
  QOL of caregivers. Two subscales of health related quality of life (QOL): physical health and mental health (score range:0-100). Higher scores indicate better QoL.
Patient Health Questionnaire - (PHQ-9; Kroenke et al., 2002) | Baseline
  Depression of caregivers. Assesses severe symptoms of depression based on criteria by the DSM IV.
  9 items, sumscore (range 0-27), a high sumscore indicates a high level of depression
Quality of Dying and Death Questionnaire for Informal Caregivers (QODD-D-Ang; Heckel et al. 2015) | 4-8 weeks after death of patient (if occuring within one year after randomisation)
  The QODD-questionnaire (Qualitiy of dying and death) assesses the quality of the deceasing phase from a caregivers perspective.QODD-D-Ang total score (sumscore range 0-100); higher scores indicate better Quality of dying and death.
Barriers of communication (caregiver) | 8 weeks; Baseline, 8 weeks (after randomisation: a.r.),
  This self developed questionnaire will try to assess the barriers of communication of patients and caregivers concerning topics like end of life care and death. The scale will be validated in the study. Higher scores indicate more barriers of communication.
Expectations about treatment of patients (self-developed, visual analogues scales) | 16 weeks; Baseline, 16 weeks (a. r.)
  These three self-developed items assess descriptive 1. the expectations caregivers have towards their relatives cancer therapy (e.g. prolonging of life, improvement of QoL) and 2. the importance of prolonging of life & improvement of QoL (two visual analogues scales)
Inventory of Complicated Grief (Lumbeck, Brandstätter, & Geissner, 2013; Prigerson et al., 1995) | 4-8 weeks after death of patient (if occuring within one year after randomisation)
  Complicated grief, 19 items, sumscore (0-76, cut-off >25)
Existence of ACP directive | 4-8 weeks after death of patient (if occuring within one year after randomisation)
  Caregivers will be asked, if the patient has completed and advance healthcare directive or took part in an ACP-process. Purely descriptive (Advance directive yes vs. no)

CONTACTS AND LOCATIONS:
Overall Officials: Carola Seifart, PD Dr. med, Principal Investigator — Philipps University Marburg; Pia von Blanckenburg, Phd., Study Director — Philipps University Marburg, Department of Psychology, Division of Clinical Psychology and Psychotherapy
Locations (2):
- Germany (2):
  - Philipps University, Departement of Psychology, Division of Clinical Psychology and Psychtherapy, Marburg
  - Philipps University, Marburg

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available after trial is finished. We have not decided to what extend and how we can provide the data.

REFERENCES:
- [Background] Ando M, Morita T, Akechi T, Okamoto T; Japanese Task Force for Spiritual Care. Efficacy of short-term life-review interviews on the spiritual well-being of terminally ill cancer patients. J Pain Symptom Manage. 2010 Jun;39(6):993-1002. doi: 10.1016/j.jpainsymman.2009.11.320. PMID 20538183
- [Background] Chochinov HM, Hack T, Hassard T, Kristjanson LJ, McClement S, Harlos M. Dignity therapy: a novel psychotherapeutic intervention for patients near the end of life. J Clin Oncol. 2005 Aug 20;23(24):5520-5. doi: 10.1200/JCO.2005.08.391. PMID 16110012
- [Background] Bollig G, Rosland JH, Gjengedal E, Schmidt G, May AT, Heller A. A European multicenter study on systematic ethics work in nursing homes. Scand J Caring Sci. 2017 Sep;31(3):587-601. doi: 10.1111/scs.12373. Epub 2016 Aug 26. PMID 27561245
- [Background] Weitzner MA, Jacobsen PB, Wagner H Jr, Friedland J, Cox C. The Caregiver Quality of Life Index-Cancer (CQOLC) scale: development and validation of an instrument to measure quality of life of the family caregiver of patients with cancer. Qual Life Res. 1999;8(1-2):55-63. doi: 10.1023/a:1026407010614. PMID 10457738
- [Background] Weitzner MA, McMillan SC. The Caregiver Quality of Life Index-Cancer (CQOLC) Scale: revalidation in a home hospice setting. J Palliat Care. 1999 Summer;15(2):13-20. PMID 10425873
- [Background] Cohen L, Parker PA, Vence L, Savary C, Kentor D, Pettaway C, Babaian R, Pisters L, Miles B, Wei Q, Wiltz L, Patel T, Radvanyi L. Presurgical stress management improves postoperative immune function in men with prostate cancer undergoing radical prostatectomy. Psychosom Med. 2011 Apr;73(3):218-25. doi: 10.1097/PSY.0b013e31820a1c26. Epub 2011 Jan 21. PMID 21257977
- [Background] Markowitz JC, Kocsis JH, Fishman B, Spielman LA, Jacobsberg LB, Frances AJ, Klerman GL, Perry SW. Treatment of depressive symptoms in human immunodeficiency virus-positive patients. Arch Gen Psychiatry. 1998 May;55(5):452-7. doi: 10.1001/archpsyc.55.5.452. PMID 9596048
- [Background] Mack JW, Nilsson M, Balboni T, Friedlander RJ, Block SD, Trice E, Prigerson HG. Peace, Equanimity, and Acceptance in the Cancer Experience (PEACE): validation of a scale to assess acceptance and struggle with terminal illness. Cancer. 2008 Jun;112(11):2509-17. doi: 10.1002/cncr.23476. PMID 18429006
- [Background] Zeng L, Bedard G, Cella D, Thavarajah N, Chen E, Zhang L, Bennett M, Peckham K, De Costa S, Beaumont JL, Tsao M, Danjoux C, Barnes E, Sahgal A, Chow E. Preliminary results of the generation of a shortened quality-of-life assessment for patients with advanced cancer: the FACIT-Pal-14. J Palliat Med. 2013 May;16(5):509-15. doi: 10.1089/jpm.2012.0595. Epub 2013 Apr 16. PMID 23590181
- [Background] Miller DC, Sanda MG, Dunn RL, Montie JE, Pimentel H, Sandler HM, McLaughlin WP, Wei JT. Long-term outcomes among localized prostate cancer survivors: health-related quality-of-life changes after radical prostatectomy, external radiation, and brachytherapy. J Clin Oncol. 2005 Apr 20;23(12):2772-80. doi: 10.1200/JCO.2005.07.116. PMID 15837992
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Heckel M, Bussmann S, Stiel S, Weber M, Ostgathe C. Validation of the German Version of the Quality of Dying and Death Questionnaire for Informal Caregivers (QODD-D-Ang). J Pain Symptom Manage. 2015 Sep;50(3):402-13. doi: 10.1016/j.jpainsymman.2015.03.020. Epub 2015 Jun 14. PMID 26079825
- [Background] Prigerson HG, Maciejewski PK, Reynolds CF 3rd, Bierhals AJ, Newsom JT, Fasiczka A, Frank E, Doman J, Miller M. Inventory of Complicated Grief: a scale to measure maladaptive symptoms of loss. Psychiatry Res. 1995 Nov 29;59(1-2):65-79. doi: 10.1016/0165-1781(95)02757-2. PMID 8771222
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Mehnert, Anja; Müller, Diana; Lehmann, Claudia; Koch, Uwe (2006): Die deutsche Version des NCCN Distress-Thermometers. In: Zeitschrift für Psychiatrie, Psychologie und Psychotherapie 54 (3), S. 213-223. DOI: 10.1024/1661-4747.54.3.213.
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Lumbeck, Gudrun; Brandstätter, Monika; Geissner, Edgar (2012): Erstvalidierung der deutschen Version des "Inventory of Complicated Grief" (ICG-D). In: Zeitschrift für Klinische Psychologie und Psychotherapie 41 (4), p. 243-248.
- [Derived] Seifart C, Koch M, Herzog S, Leppin N, Nagelschmidt K, Riera Knorrenschild J, Timmesfeld N, Denz R, Seifart U, Rief W, Von Blanckenburg P. Collaborative advance care planning in palliative care: a randomised controlled trial. BMJ Support Palliat Care. 2024 Jul 2:spcare-2023-004175. doi: 10.1136/spcare-2023-004175. Online ahead of print. PMID 38960600
- [Derived] Seifart C, Koch M, Leppin N, Nagelschmidt K, Knorrenschild JR, Timmesfeld N, Rief W, von Blanckenburg P. Collaborative advance care planning in advanced cancer patients: col-ACP -study - study protocol of a randomised controlled trial. BMC Palliat Care. 2020 Aug 24;19(1):134. doi: 10.1186/s12904-020-00629-7. PMID 32838763